CLINICAL TRIAL: NCT01661998
Title: Motion Preservation Evaluation Below Fusions of the Spine in Adolescent Idiopathic Scoliosis
Brief Title: Prospective Study of Motion Preservation Evaluation Below Fusions of the Spine in Adolescent Idiopathic Scoliosis
Acronym: POM
Status: Completed | Type: Observational
Sponsor: Setting Scoliosis Straight Foundation (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009HSGF05
Record Dates: First submitted 2012-07-10; First posted 2012-08-10 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2019-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Spinal Deformity; Treatment Outcomes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Harms Study Group

SUMMARY:
The purpose of this study is to evaluate the relationship of A) The distal fusion level B) The total length of fusion and the post-operative range of motion in the unfused vertebral segments below the fusion in patients with Adolescent Idiopathic Scoliosis.

DETAILED DESCRIPTION:
The motion behavior in the unfused segments of the spine following instrumentation is poorly understood and the implications of hyper or hypo-mobility have not been clearly defined. The purpose of this study is to evaluate the relationship of A) The distal fusion level B) The total length of fusion and the post-operative range of motion in the unfused vertebral segments below the fusion in patients with Adolescent Idiopathic Scoliosis to answer the following specific clinical questions:

1. Further elucidate the motion behavior of the distal unfused spinal segments, specifically:

   1. Does motion differ at various post-operative time points (2 year post-op patients versus 5 or 10 year post-op patients)?
   2. Can predictive factors be identified with post-operative altered motion?
2. Further elucidate the relationship of the motion in the unfused spinal segments to the lowest instrumented vertebrae.
3. Determine the relationship of the total length of fusion to the motion in the unfused spinal segments (i.e. compare unfused motion in the distal unfused segments in Lenke 5/6 patients fused selectively (ThL/L only) versus nonselectively (TH and ThL/L)).
4. Determine the relationship between clinical examinations (i.e. reports of pain or functional limitations) and patient reported outcomes (Health Related Quality of Life Outcome Tools) to motion in the distal unfused segments.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the primary and co-investigator's facilities will be offered inclusion into the study if they meet the following inclusion criteria:

  * Patient age < 21 years
  * Male or female
  * Diagnosis of Adolescent Idiopathic Scoliosis
  * Any Lenke Classification type
  * Underwent surgical correction of the spinal deformity with a fusion
  * Are due for their 10 year post-operative visit

Exclusion Criteria:

* Patients will be excluded from study inclusion if they meet the following exclusion criteria:

  * Neuromuscular co-morbidity

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who present to the investigator's clinic, who meet the inclusion criteria will be offered enrollment in the study
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2008-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Evaluate post-operative range of motion in the unfused vertebral segments below the fusion in patients with Adolescent Idiopathic Scoliosis. Range of motion is assessed by side-bending to the left and to the right as well as bending forward. | 10 years
  Data collected at patients 10 years visit.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Newton, MD, Study Director — Rady Children's Hospital San Deigo
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - Scoliosis Associates & NYU Hospital for Joint Diseases, New York, New York
  - Shriners Hospital for Children, Philadelphia, Pennsylvania

REFERENCES:
- See also: Setting Scoliosis Straight Website - highlighting the research of the Harms Study Group — http://hsg.settingscoliosisstraight.org/current-hsg-research/